CLINICAL TRIAL: NCT00855946
Title: Proteomic Approach Using Matrix-assisted Laser Desorption/Ionization Tandem Time-of-flight (MALDI-TOF/TOF) of Tumor Response in Rectal Carcinoma After Radiochemotherapy
Acronym: PROTEORECTUM
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX - 2008/25
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Rectal Adenocarcinoma
Keywords: tumor response; rectal adenocarcinoma; preoperative radiochemotherapy; Proteomic analysis; MALDI-TOF-TOF; rectal adenocarcinoma, tumor response after preoperative radiochemotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Treatment for locally-advanced rectal adenocarcinoma includes preoperative radiochemotherapy before surgery with total mesorectal excision in order to reduce tumor infiltration, facilitate oncologic surgery and improve survival. About fifty percent of these patients are good responders i.e. their tumor infiltration reduces in the rectal wall and regional lymph nodes in order to be graded ypT0 to T2 N0 after pathologic assessment (so called downstaging). At the opposite, bad responders (ypT3-4 and/or N+) are not sensitive to standard preoperative radiochemotherapy, and their survival is poor than good responders. Until now, response to preoperative radiochemotherapy cannot be anticipated before pathological assessment of surgical specimen. Proteomic analysis of sera from good and bad responders to preoperative radiochemotherapy could allow identification of early biomarkers of tumor response, and subsequently adaptation of treatment to increase preoperative treatment efficiency and survival in most patients.

DETAILED DESCRIPTION:
Good or bad responders to preoperative radiochemotherapy for locally-advanced rectal adenocarcinoma cannot be anticipated before pathological assessment of rectal specimen. The purpose of this prospective monocentric study is to look for early seric biomarkers predictive of tumor response (good and bad responders) in patients treated by preoperative radiochemotherapy (45 Gy) for rectal adenocarcinoma using a proteomic approach. All patients with locally-advanced rectal adenocarcinoma will be enrolled. Sequential samples of sera will be collected before, during preoperative treatment and before surgery, and analysed using a MALDI-TOF-TOF method. Proteomic analysis will be correlated to pathological response in order to identify potential early biomarkers of tumor response.

ELIGIBILITY:
Inclusion Criteria:

* T3T4 or N+ M0 rectal carcinoma
* histologically-proven adenocarcinoma
* from 0 to 15 cm from the anal verge
* patient is at least 18 years of age
* ECOG performance status </= 2
* Patient and doctor have signed informed consent

Exclusion Criteria:

* Metastatic disease
* T1-T2 N0 rectal carcinoma
* Contra indication of radiotherapy or chemotherapy
* History of cancer
* Severe renal insufficiency
* Symptomatic cardiac or coronary insufficiency
* Patient included in a trial
* Previous radiotherapy or chemotherapy for this cancer
* No contraceptive treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with rectal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
differential expression of early seric biomarkers between good and bad responders. | at inclusion and 24-48h after starting radiochemotherapy

SECONDARY OUTCOMES:
modifications of isolated biomarkers within presurgical period | at inclusion, 24-48h after initiation of radiochemotherapy, at the end of radiochemotherapy (6th week) and before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne RULLIER, MD, Principal Investigator — University Hospital Bordeaux, France; Paul PEREZ, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Laboratoire d'anatomie pathologique, University Hospital, Bordeaux, Bordeaux, France

REFERENCES:
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] Kapiteijn E, Marijnen CA, Nagtegaal ID, Putter H, Steup WH, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van Krieken JH, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med. 2001 Aug 30;345(9):638-46. doi: 10.1056/NEJMoa010580. PMID 11547717
- [Background] Pahlman L, Glimelius B. Radiotherapy additional to surgery in the management of primary rectal carcinoma. Acta Chir Scand. 1990 Jun-Jul;156(6-7):475-85. No abstract available. PMID 2195818
- [Background] Swedish Rectal Cancer Trial; Cedermark B, Dahlberg M, Glimelius B, Pahlman L, Rutqvist LE, Wilking N. Improved survival with preoperative radiotherapy in resectable rectal cancer. N Engl J Med. 1997 Apr 3;336(14):980-7. doi: 10.1056/NEJM199704033361402. PMID 9091798
- [Background] Randomised trial of surgery alone versus radiotherapy followed by surgery for potentially operable locally advanced rectal cancer. Medical Research Council Rectal Cancer Working Party. Lancet. 1996 Dec 14;348(9042):1605-10. PMID 8961989
- [Background] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Bosset JF, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Briffaux A, Collette L. Enhanced tumorocidal effect of chemotherapy with preoperative radiotherapy for rectal cancer: preliminary results--EORTC 22921. J Clin Oncol. 2005 Aug 20;23(24):5620-7. doi: 10.1200/JCO.2005.02.113. Epub 2005 Jul 11. PMID 16009958
- [Background] Vecchio FM, Valentini V, Minsky BD, Padula GD, Venkatraman ES, Balducci M, Micciche F, Ricci R, Morganti AG, Gambacorta MA, Maurizi F, Coco C. The relationship of pathologic tumor regression grade (TRG) and outcomes after preoperative therapy in rectal cancer. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):752-60. doi: 10.1016/j.ijrobp.2004.11.017. PMID 15936556
- [Background] Rodel C, Martus P, Papadoupolos T, Fuzesi L, Klimpfinger M, Fietkau R, Liersch T, Hohenberger W, Raab R, Sauer R, Wittekind C. Prognostic significance of tumor regression after preoperative chemoradiotherapy for rectal cancer. J Clin Oncol. 2005 Dec 1;23(34):8688-96. doi: 10.1200/JCO.2005.02.1329. Epub 2005 Oct 24. PMID 16246976
- [Background] Garcia-Aguilar J, Hernandez de Anda E, Sirivongs P, Lee SH, Madoff RD, Rothenberger DA. A pathologic complete response to preoperative chemoradiation is associated with lower local recurrence and improved survival in rectal cancer patients treated by mesorectal excision. Dis Colon Rectum. 2003 Mar;46(3):298-304. doi: 10.1007/s10350-004-6545-x. PMID 12626903
- [Background] Moore HG, Gittleman AE, Minsky BD, Wong D, Paty PB, Weiser M, Temple L, Saltz L, Shia J, Guillem JG. Rate of pathologic complete response with increased interval between preoperative combined modality therapy and rectal cancer resection. Dis Colon Rectum. 2004 Mar;47(3):279-86. doi: 10.1007/s10350-003-0062-1. PMID 14991488
- [Background] Collette L, Bosset JF, den Dulk M, Nguyen F, Mineur L, Maingon P, Radosevic-Jelic L, Pierart M, Calais G; European Organisation for Research and Treatment of Cancer Radiation Oncology Group. Patients with curative resection of cT3-4 rectal cancer after preoperative radiotherapy or radiochemotherapy: does anybody benefit from adjuvant fluorouracil-based chemotherapy? A trial of the European Organisation for Research and Treatment of Cancer Radiation Oncology Group. J Clin Oncol. 2007 Oct 1;25(28):4379-86. doi: 10.1200/JCO.2007.11.9685. PMID 17906203
- [Background] Habr-Gama A, Perez RO, Nadalin W, Nahas SC, Ribeiro U Jr, Silva E Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Long-term results of preoperative chemoradiation for distal rectal cancer correlation between final stage and survival. J Gastrointest Surg. 2005 Jan;9(1):90-9; discussion 99-101. doi: 10.1016/j.gassur.2004.10.010. PMID 15623449
- [Background] Peeters KC, van de Velde CJ, Leer JW, Martijn H, Junggeburt JM, Kranenbarg EK, Steup WH, Wiggers T, Rutten HJ, Marijnen CA. Late side effects of short-course preoperative radiotherapy combined with total mesorectal excision for rectal cancer: increased bowel dysfunction in irradiated patients--a Dutch colorectal cancer group study. J Clin Oncol. 2005 Sep 1;23(25):6199-206. doi: 10.1200/JCO.2005.14.779. PMID 16135487
- [Background] Murata A, Brown CJ, Raval M, Phang PT. Impact of short-course radiotherapy and low anterior resection on quality of life and bowel function in primary rectal cancer. Am J Surg. 2008 May;195(5):611-5; discussion 615. doi: 10.1016/j.amjsurg.2007.12.034. PMID 18367144
- [Background] Pollack J, Holm T, Cedermark B, Holmstrom B, Mellgren A. Long-term effect of preoperative radiation therapy on anorectal function. Dis Colon Rectum. 2006 Mar;49(3):345-52. doi: 10.1007/s10350-005-0296-1. PMID 16532369
- [Background] Lopez-Crapez E, Bibeau F, Thezenas S, Ychou M, Simony-Lafontaine J, Thirion A, Azria D, Grenier J, Senesse P. p53 status and response to radiotherapy in rectal cancer: a prospective multilevel analysis. Br J Cancer. 2005 Jun 20;92(12):2114-21. doi: 10.1038/sj.bjc.6602622. PMID 15956964
- [Background] Gunther K, Dimmler A, Rodel F, Reulbach U, Merkel S, Bittorf BR, Matzel KE, Papadopoulos T, Hohenberger W, Sauer R, Rodel C. P27 does not predict histopathological response to radiochemotherapy in rectal cancer. J Surg Res. 2003 Aug;113(2):179-88. doi: 10.1016/s0022-4804(03)00049-0. PMID 12957127
- [Background] Rau B, Sturm I, Lage H, Berger S, Schneider U, Hauptmann S, Wust P, Riess H, Schlag PM, Dorken B, Daniel PT. Dynamic expression profile of p21WAF1/CIP1 and Ki-67 predicts survival in rectal carcinoma treated with preoperative radiochemotherapy. J Clin Oncol. 2003 Sep 15;21(18):3391-401. doi: 10.1200/JCO.2003.07.077. Epub 2003 Jul 28. PMID 12885834
- [Background] Komuro Y, Watanabe T, Tsurita G, Muto T, Nagawa H. Evaluating the combination of molecular prognostic factors in tumor radiosensitivity in rectal cancer. Hepatogastroenterology. 2005 May-Jun;52(63):666-71. PMID 15966178
- [Background] Smith FM, Reynolds JV, Miller N, Stephens RB, Kennedy MJ. Pathological and molecular predictors of the response of rectal cancer to neoadjuvant radiochemotherapy. Eur J Surg Oncol. 2006 Feb;32(1):55-64. doi: 10.1016/j.ejso.2005.09.010. Epub 2005 Dec 1. PMID 16324817
- [Background] Barratt PL, Seymour MT, Stenning SP, Georgiades I, Walker C, Birbeck K, Quirke P; UKCCCR AXIS trial collaborators. Adjuvant X-ray and Fluorouracil Infusion Study. DNA markers predicting benefit from adjuvant fluorouracil in patients with colon cancer: a molecular study. Lancet. 2002 Nov 2;360(9343):1381-91. doi: 10.1016/s0140-6736(02)11402-4. PMID 12423985
- [Background] Giralt J, Eraso A, Armengol M, Rossello J, Majo J, Ares C, Espin E, Benavente S, de Torres I. Epidermal growth factor receptor is a predictor of tumor response in locally advanced rectal cancer patients treated with preoperative radiotherapy. Int J Radiat Oncol Biol Phys. 2002 Dec 1;54(5):1460-5. doi: 10.1016/s0360-3016(02)03752-5. PMID 12459370
- [Background] Smith FM, Reynolds JV, Kay EW, Crotty P, Murphy JO, Hollywood D, Gaffney EF, Stephens RB, Kennedy MJ. COX-2 overexpression in pretreatment biopsies predicts response of rectal cancers to neoadjuvant radiochemotherapy. Int J Radiat Oncol Biol Phys. 2006 Feb 1;64(2):466-72. doi: 10.1016/j.ijrobp.2005.07.961. Epub 2005 Oct 5. PMID 16213106
- [Background] Komuro Y, Watanabe T, Hosoi Y, Matsumoto Y, Nakagawa K, Tsuno N, Kazama S, Kitayama J, Suzuki N, Nagawa H. The expression pattern of Ku correlates with tumor radiosensitivity and disease free survival in patients with rectal carcinoma. Cancer. 2002 Sep 15;95(6):1199-205. doi: 10.1002/cncr.10807. PMID 12216085
- [Background] Rodel F, Hoffmann J, Distel L, Herrmann M, Noisternig T, Papadopoulos T, Sauer R, Rodel C. Survivin as a radioresistance factor, and prognostic and therapeutic target for radiotherapy in rectal cancer. Cancer Res. 2005 Jun 1;65(11):4881-7. doi: 10.1158/0008-5472.CAN-04-3028. PMID 15930309
- [Background] Milas L, Mason KA, Ariga H, Hunter N, Neal R, Valdecanas D, Krieg AM, Whisnant JK. CpG oligodeoxynucleotide enhances tumor response to radiation. Cancer Res. 2004 Aug 1;64(15):5074-7. doi: 10.1158/0008-5472.CAN-04-0926. PMID 15289307
- [Background] Rodel C, Grabenbauer GG, Papadopoulos T, Bigalke M, Gunther K, Schick C, Peters A, Sauer R, Rodel F. Apoptosis as a cellular predictor for histopathologic response to neoadjuvant radiochemotherapy in patients with rectal cancer. Int J Radiat Oncol Biol Phys. 2002 Feb 1;52(2):294-303. doi: 10.1016/s0360-3016(01)02643-8. PMID 11872273
- [Background] Ghadimi BM, Grade M, Difilippantonio MJ, Varma S, Simon R, Montagna C, Fuzesi L, Langer C, Becker H, Liersch T, Ried T. Effectiveness of gene expression profiling for response prediction of rectal adenocarcinomas to preoperative chemoradiotherapy. J Clin Oncol. 2005 Mar 20;23(9):1826-38. doi: 10.1200/JCO.2005.00.406. PMID 15774776
- [Background] Smith FM, Gallagher WM, Fox E, Stephens RB, Rexhepaj E, Petricoin EF 3rd, Liotta L, Kennedy MJ, Reynolds JV. Combination of SELDI-TOF-MS and data mining provides early-stage response prediction for rectal tumors undergoing multimodal neoadjuvant therapy. Ann Surg. 2007 Feb;245(2):259-66. doi: 10.1097/01.sla.0000245577.68151.bd. PMID 17245180
- [Background] Hudelist G, Singer CF, Pischinger KI, Kaserer K, Manavi M, Kubista E, Czerwenka KF. Proteomic analysis in human breast cancer: identification of a characteristic protein expression profile of malignant breast epithelium. Proteomics. 2006 Mar;6(6):1989-2002. doi: 10.1002/pmic.200500129. PMID 16470630
- [Background] Le Moguen K, Lincet H, Marcelo P, Lemoisson E, Heutte N, Duval M, Poulain L, Vinh J, Gauduchon P, Baudin B. A proteomic kinetic analysis of IGROV1 ovarian carcinoma cell line response to cisplatin treatment. Proteomics. 2007 Nov;7(22):4090-101. doi: 10.1002/pmic.200700231. PMID 17994630